CLINICAL TRIAL: NCT06016127
Title: A Single-center, Randomized, Pilot Study to Assess Iovera° Lumbar Medial Branch Cryoneurolysis vs Lumbar Radiofrequency Ablation for Facet Mediated Chronic Low Back Pain
Brief Title: Cryoneurolysis for Facet Mediated Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Pain Management Services, PLLC (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRS-107
Record Dates: First submitted 2023-08-21; First posted 2023-08-29 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Low Back Pain; Facet Joint Pain
Keywords: low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Randomization to treatment groups according to the randomization assignment
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cryoneurolysis (Active Comparator): Subjects will receive iovera° cryoneurolysis to the medial branch nerves of the lumbar spine
  Interventions: Device: iovera system
- Radiofrequency ablation (Active Comparator): Subjects will receive RFA to the medial branch nerves of the lumbar spine
  Interventions: Device: Radiofrequency ablation

INTERVENTIONS:
Device: iovera system — The iovera° system consists of a reusable, portable Handpiece, along with single patient use sterile Smart Tips (i.e., cryoprobes) and disposable nitrous oxide (N2O) cartridges. The iovera° system produces the desired effect through initiation of a cooling cycle. Each cooling cycle is initiated by fully inserting the Smart Tip into the selected procedure site and activating the cryogen flow. The Smart Tip needles are made of stainless steel and have a closed tip, fully enclosing the cryogen. The "190" Smart Tip will be used in this study.
  Other Names: iovera
  Arms: Cryoneurolysis
Device: Radiofrequency ablation — The RFA system consists of a Cosman, G4 Generator. The needles used are 20-gauge, 10cm long with a 10mm active tip manufactured by Cosman. A grounding pad, also manufactured by Cosman, is placed on the upper thigh for each procedure and connected to the G4 Generator.
  Arms: Radiofrequency ablation

SUMMARY:
This is a single-center, randomized, pilot study in adult subjects with facet mediated CLBP. Thirty (30) subjects are planned for initial enrollment and will be randomized 1:1 to receive ioveraº medial branch cryoneurolysis or radiofrequency ablation.

DETAILED DESCRIPTION:
This is a single-center, randomized, pilot study in adult subjects with facet mediated CLBP. Thirty (30) subjects are planned for initial enrollment and will be randomized 1:1 to receive ioveraº medial branch cryoneurolysis or radiofrequency ablation.

This study is designed to determine if a full efficacy RCT can be successfully conducted using the procedures and protocols described in the current pilot study protocol, or if protocol modifications are necessary before moving forward with a full efficacy RCT. Furthermore, the study will assess the feasibility of the outcome measurements employed, construct a foundation for sample size calculation, and the acceptability/practicality of conducting the full efficacy RCT.

Randomization to treatment groups according to the randomization assignment will be performed on the day of treatment. The treatment groups are:

* Group 1: subjects will receive iovera° cryoneurolysis to the medial branch nerves of the lumbar spine
* Group 2: subjects will receive RFA to the medial branch nerves of the lumbar spine

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers, at least 18 years of age at screening
2. Primary complaint of axial low-back pain suggestive of unilateral or bilateral facet joint involvement (i.e., facet mediated CLBP)
3. Low back pain is chronic (i.e., > 3 months' duration)
4. Low back pain score of ≥ 4 (i.e., moderate pain) on the 0 to 10 NRS or functional impairment at screening
5. Successful trial of two diagnostic medial branch blocks consisting of two positive blocks with local anesthetic only (i.e., no steroids) that results in at least 50% relief of primary (index) pain for the duration of the local anesthetic used or history of a positive response to prior radiofrequency treatment (i.e., ≥ 6 months prior to enrollment)
6. Failure of at least three months of conservative non-operative therapy (e.g., physical therapy, chiropractic care, spinal injections, NSAIDs or other appropriate analgesics),
7. Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments

Exclusion Criteria:

1. Active workers' compensation, personal injury, Social Security disability insurance (SSDI), or other litigation/compensation related to the spine
2. Serious spinal disorders (verified on magnetic resonance imaging (MRI)) that may impact outcomes, including any of the following:

   1. Suspected cauda equina syndrome (e.g., bowel/bladder dysfunction)
   2. Infection
   3. Tumor
   4. Traumatic fracture
   5. Systemic inflammatory spondyloarthropathy
   6. Lumbar radiculopathy/radiculitis (i.e., root irritation and deficit)
   7. Neurogenic claudication
3. Prior lumbar spinal fusion surgery
4. Comorbidity that, in the judgment of the Investigator, may affect the subject's ability to participate in the study including lumbar radiculopathy and neuropathic pain disorder
5. Currently pregnant, nursing, or planning to become pregnant during the study
6. Known contraindication to study devices, including any of the following:

   1. Cryoglobulinemia
   2. Paroxysmal cold hemoglobinuria
   3. Cold urticaria
   4. Raynaud's disease
   5. Open and/or infected wounds at or near the treatment site
   6. Coagulopathy
7. 3.5-inch needle cannot be used in the low back region because of habitus
8. Severe chronic pain disorder that in the opinion of the investigator may impact postsurgical outcomes
9. Presence of any of the following:

   1. Spinal neurostimulator
   2. Intrathecal analgesic drug pump
10. Current manifestation of poorly controlled mental illness that in the opinion of the investigator may meaningfully impact treatment outcomes, including any of the following:

    1. Mood disorder (e.g., major depression, bipolar)
    2. Psychotic disorder (e.g., schizophrenia)
11. Subject received other spine intervention/therapies in the 30 days prior to block administration (e.g., spinal injections, minimally invasive therapies, surgical therapies)
12. Subject received radiofrequency ablation in the low back region ≤ 6 months before study enrollment
13. History, suspicion, or clinical manifestation of:

    1. Alcohol abuse or dependence
    2. Illicit drug use
    3. Opioid abuse or dependence (≥40 mg MED PO/day in past 30 days) Given the COVID-19 pandemic, the subject must be medically fit/cleared for treatment by the investigator. If there is a concern about a subject's recent or potential exposure to COVID-19, or if the subject is not medically fit/cleared for treatment due to suspected COVID-19 illness/symptoms (or other serious illness), the subject must be excluded per Exclusion criterion #4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-18 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Albany & Saratoga Centers For Pain Management, Saratoga Springs, New York, United States

IPD SHARING:
Plan to Share IPD: No
Contact PI

RESULTS

PARTICIPANT FLOW:
Groups:
- Cryoneurolysis: Subjects received iovera° cryoneurolysis to the medial branch nerves of the lumbar spine
  iovera system: The iovera° system consists of a reusable, portable Handpiece, along with single patient use sterile Smart Tips (i.e., cryoprobes) and disposable nitrous oxide (N2O) cartridges. The iovera° system produces the desired effect through initiation of a cooling cycle. Each cooling cycle is initiated by fully inserting the Smart Tip into the selected procedure site and activating the cryogen flow. The Smart Tip needles are made of stainless steel and have a closed tip, fully enclosing the cryogen. The "190" Smart Tip will be used in this study.
- Radiofrequency Ablation: Subjects received RFA to the medial branch nerves of the lumbar spine
  Radiofrequency ablation: The RFA system consists of a Cosman, G4 Generator. The needles used are 20-gauge, 10cm long with a 10mm active tip manufactured by Cosman. A grounding pad, also manufactured by Cosman, is placed on the upper thigh for each procedure and connected to the G4 Generator.
Period: Overall Study
Arm/Group | Cryoneurolysis | Radiofrequency Ablation
Started | 15 | 15
Completed | 11 | 12
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Cryoneurolysis: The iovera° system consists of a reusable, portable Handpiece, along with single patient use sterile Smart Tips (i.e., cryoprobes) and disposable nitrous oxide (N2O) cartridges. The iovera° system produces the desired effect through initiation of a cooling cycle. Each cooling cycle is initiated by fully inserting the Smart Tip into the selected procedure site and activating the cryogen flow. The Smart Tip needles are made of stainless steel and have a closed tip, fully enclosing the cryogen. The "190" Smart Tip was used in this study.
- Radiofrequency Ablation: The RFA system consisted of a Cosman, G4 Generator. The needles used were 20-gauge, 10cm long with a 10mm active tip manufactured by Cosman. A grounding pad, also manufactured by Cosman was placed on the upper thigh for each procedure and connected to the G4 Generator.
- Total: Total of all reporting groups
Arm/Group | Cryoneurolysis | Radiofrequency Ablation | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (17.1) | 63.1 (12.7) | 64.5 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
NRS [Mean (Standard Deviation); unit: units on a scale] — Subjects will evaluate their pain in the low back region using an 11-point Numeric Rating Scale (NRS), where 0=no pain and 10=worst possible pain.
  Subjects will evaluate how much pain they are currently experiencing and their average pain level over the past 24 hours.
  units on a scale | 6.1 (1.8) | 6.1 (1.9) | 6.1 (1.9)
ODI [Mean (Standard Deviation); unit: units on a scale] — Function disability will be measured by the Oswestry Disability Index. The score ranges from 0-50, with lower scores reflecting milder disability.
  units on a scale | 18.5 (7.1) | 18.7 (5.9) | 18.6 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Safety of Cryoneurolysis as Compared to Radiofrequency Ablation (RFA)
Description: Safety will be assessed as the number of subjects with reported treatment-related adverse related to cryoneurolysis or RFA.
Time Frame: 0-12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoneurolysis | Radiofrequency Ablation
Number analyzed (Participants) | 11 | 12
Participants | 0 | 0

2. Secondary Outcome: Pain Intensity as Measured by 11-point Numeric Rating Scale (NRS) at 12 Month Follow up
Description: Subjects will evaluate their pain in the low back region using an 11-point Numeric Rating Scale (NRS), where 0=no pain and 10=worst possible pain.
  Subjects will evaluate how much pain they are currently experiencing and their average pain level over the past 24 hours.
Time Frame: 12 months
Population: Subjects who received the study intervention and completed 12-month study follow-up.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cryoneurolysis | Radiofrequency Ablation
Number analyzed (Participants) | 11 | 12
units on a scale | 3.04 (0.77) | 6.13 (0.77)

3. Other Pre Specified Outcome: Functional Disability Index at 12 Month Follow up
Description: Function disability will be measured by the Oswestry Disability Index. The score ranges from 0-50, with lower scores reflecting milder disability.
Time Frame: 0-12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cryoneurolysis | Radiofrequency Ablation
Number analyzed (Participants) | 11 | 12
score on a scale | 10.15 [6.00 to 14.30] | 20.61 [16.47 to 24.74]

4. Other Pre Specified Outcome: Patients' Global Impression of Change at 12 Month Follow up
Description: The Patients' Global Impression of Change (PGIC) is an 11-point self-report scale assessing overall changes in activity limitations, symptoms, emotions, and quality of life, ranging from 0 to 10, where higher values indicate worse outcomes.
Time Frame: 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cryoneurolysis | Radiofrequency Ablation
Number analyzed (Participants) | 11 | 12
score on a scale | 1.74 [0.70 to 2.77] | 4.38 [3.34 to 5.41]

5. Other Pre Specified Outcome: Satisfaction With Pain Management
Description: Subject satisfaction with pain management as measured on a scale ranging from 1) extremely dissatisfied 2) dissatisfied 3) neither satisfied nor dissatisfied 4) satisfied 5) extremely satisfied.
Time Frame: 12 months
Population: Subjects who received the study intervention and completed the 12-month follow-up.
Measure: Number; unit: participants
Arm/Group | Cryoneurolysis | Radiofrequency Ablation
Number analyzed (Participants) | 11 | 12
participants
  Dissatisfied | 0 | 0
  Neither satisfied nor dissatisfied | 1 | 4
  Satisfied | 10 | 8

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cryoneurolysis | Radiofrequency Ablation
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryoneurolysis (N=15) | Radiofrequency Ablation (N=15)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT06016127/Prot_002.pdf
  • Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT06016127/SAP_003.pdf